CLINICAL TRIAL: NCT06484868
Title: A 24-Month, Multi-Centre, Open Label Phase IV Post Authorisation Efficacy Study to Evaluate the Efficacy, Safety and Immunogenicity of Daily Subcutaneous Metreleptin Treatment in Patients With Partial Lipodystrophy
Brief Title: Open-label Study to Evaluate Metreleptin in Patients With Partial Lipodystrophy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amryt Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL-22; 2022-502950-14-00 (EU CTIS Number)
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Partial Lipodystrophy
Keywords: Metreleptin
MeSH Terms: conditions — Lipodystrophy, Partial, Acquired | interventions — metreleptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metreleptin (Experimental): Metreleptin [Recombinant-methionyl human Leptin; r-metHuLeptin] for daily injection is a sterile, white, solid lyophilised cake
  Interventions: Drug: Metreleptin

INTERVENTIONS:
Drug: Metreleptin — Metreleptin is a recombinant human leptin analog that is indicated as an adjunct to diet as replacement therapy to treat the complications of leptin deficiency

SUMMARY:
This is an Open Label, Phase IV, Post Authorisation Study to Evaluate the Efficacy, Safety and Immunogenicity of Daily Subcutaneous Metreleptin Treatment in people with Partial Lipodystrophy

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of familial or acquired partial lipodystrophy

Exclusion Criteria:

* Treatment with any Investigational Medicinal Product (IMP) within 6 months or 5 times the terminal half-life of the corresponding IMP, whichever is longer, before the screening visit.

Other protocol defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients with decrease of at least 0.5% in glycated haemoglobin (HbA1c) at Month 12 compared to Baseline or HbA1c <6.5 % at Month 12, in patients with baseline HbA1c ≥6.5%. | 12 months
  To evaluate the efficacy (HbA1c) of metreleptin treatment in patients with PL
Number of patients with decrease of at least 30% in triglycerides (TG) at Month 12 compared to Baseline, in patients with baseline TG levels ≥500 mg/dL (5.65 mmol/L) | 12 months
  To evaluate the efficacy (TG) of metreleptin treatment in patients with PL

SECONDARY OUTCOMES:
Number of patients with decrease of at least 0.5% in HbA1c at Month 24 compared to Baseline or HbA1c <6.5 % at Month 24, in patients with baseline HbA1c ≥6.5%. | 24 months
  To evaluate the long-term efficacy of metreleptin treatment in patients with PL
Number of patients with decrease of at least 30% in TG levels at Month 24 compared to Baseline, in patients with baseline TG levels ≥500 mg/dL (5.65 mmol/L). | 24 months
  To evaluate the long-term efficacy of metreleptin treatment in patients with PL
Change from baseline in liver volume at Month 12 and Month 24 | 12 months and 24 months
  To assess changes in liver volume.
Incidence of, Treatment emergent adverse events (TEAEs), Deaths and other serious adverse events (SAEs), Treatment related adverse events (AEs), AEs of special interest (AESIs) and AEs leading to study drug discontinuation | 24 months
  To evaluate the safety of metreleptin treatment in patients with PL

CONTACTS AND LOCATIONS:
Locations (12):
- France (4):
  - Centre Hospitalier Régional Universitaire de Lille (CHRU) - Hôpital Claude Huriez, Lille
  - Hopital Pitie-Salpetriere, Paris
  - Hôpital Saint-Antoine, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (2):
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Universitaetsklinikum Ulm - Klinik fuer Kinder- und Jugendmedizin, Ulm
- Italy (5):
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna
  - Universitá degli Studi "Magna Graecia" di Catanzaro, Catanzaro
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Novara
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
  - A.S.U Integrata di Udine - Presidio Ospedaliero Santa Maria della Misericordia, Udine
- Cambridge University Hospitals NHS Foundation Trust - Addenbrookes Hospital, Cambridge, United Kingdom